CLINICAL TRIAL: NCT01077310
Title: Alcohol Pharmacotherapy for HIV+ Prisoners With Alcohol Dependence and Problem Drinking
Brief Title: Alcohol Pharmacotherapy for HIV+ Prisoners
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0908005572; 1R01AA018944 (NIH)
Record Dates: First submitted 2010-02-19; First posted 2010-03-01 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Alcohol Dependence; Problem Drinking; Hazardous Drinking; Human Immunodeficiency Virus; AIDS
Keywords: HIV; Acquired Immunodeficiency Syndrome; Alcohol dependence; CD4; HIV-1 RNA; Alcohol treatment outcomes
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome | interventions — vivitrol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramuscular naltrexone (Active Comparator): Subjects in this arm will receive monthly intramuscular gluteal injections of depot naltrexone 380mg (VIVITROL) for 6 months. The 1st injection will be administered prior to release from prison or jail.
  Interventions: Drug: Vivitrol- Intramuscular naltrexone (depot-formulation)
- Placebo (Placebo Comparator): Subjects in this arm will receive monthly intramuscular gluteal injections of placebo for 6 months. The 1st injection will be administered prior to release from prison or jail.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vivitrol- Intramuscular naltrexone (depot-formulation) — Subjects in this arm will receive monthly intramuscular gluteal injections of depot naltrexone 380mg (VIVITROL) for 6 months. The 1st injection will be administered prior to release from prison or jail.
  Other Names: VIVITROL; extended release naltrexone; Intramuscular naltrexone; Depot-naltrexone
  Arms: Intramuscular naltrexone
Drug: Placebo — Subjects in this arm will receive monthly intramuscular gluteal injections of placebo for 6 months. The 1st injection will be administered prior to release from prison or jail. Placebo will be provided by Alkermes pharmaceuticals, the manufacturer of VIVITROL. Placebo will be identical in shape and form to active drug.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial of injectable intramuscular naltrexone (XR-NTX) versus intramuscular placebo among HIV-infected prisoners meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for alcohol dependence or problem drinking, who are transitioning to the community and seeking treatment to prevent relapse to alcohol use. We hypothesize that extended release naltrexone (XR-NTX) will result in improved HIV outcomes (lower log10 HIV-1RNA levels and higher CD4 count) as well as improved alcohol treatment outcomes, and reduced drug/sex HIV related risk behaviors and decreased rates of reincarceration.

DETAILED DESCRIPTION:
INSPIRE is a randomized controlled trial of injectable intramuscular NTX (XR-NTX) versus intramuscular placebo among Human Immunodeficiency (HIV) infected prisoners meeting DSM-IV criteria for alcohol dependence or problem drinking, who are transitioning to the community and seeking treatment to prevent relapse to alcohol use. While the COMBINE trial has demonstrated the effectiveness of oral naltrexone in a group of active alcohol dependent persons in decreasing relapse to alcohol use over placebo, naltrexone has not been studied in people who have a history of current alcohol dependence prior to incarceration, are incarcerated and not actively using alcohol and are likely to return to alcohol use when released. In this study, we conduct a placebo-controlled trial to determine if naltrexone has an effect in this group, which could be important in making the case for having naltrexone available to alcohol dependent or problem drinking HIV+ prisoners prior to release. We will compare their HIV treatment (HIV-1 RNA levels, CD4 count), alcohol treatment (time to relapse to heavy drinking, percent of days drinking, percent of days abstinent and alcohol craving) and HIV risk behavior (sexual and drug-related risks) outcomes. The hypotheses include:

i. XR-NTX will result in improved HIV clinical outcomes, including changes in HIV-1 RNA levels, and higher CD4 counts.

ii. XR-NTX will result in improved alcohol treatment outcomes, including longer time to alcohol relapse, lower percent days drinking, and lower craving for alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+
2. Inmates returning to New Haven or Hartford
3. Meets criteria for alcohol dependence (using Diagnostic and Statistical Manual IV) or problem drinking (using Alcohol Use Disorder Identification Test-AUDIT)
4. Gives informed consent
5. English or Spanish speaker
6. > 18 yrs

Exclusion Criteria:

1. On opiate pain medication or expressing need for them
2. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) > 5x the upper limit of normal
3. Evidence of Child's Pugh Class C cirrhosis
4. Pending felony charges
5. Pregnant or unwilling to take contraceptive measures
6. Subject is part of another pharmacological research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Springer, MD, Principal Investigator — Yale University; Frederick L Altice, MD, Principal Investigator — Yale University
Locations (1):
- Yale Clinical Research, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Springer SA, Altice FL, Herme M, Di Paola A. Design and methods of a double blind randomized placebo-controlled trial of extended-release naltrexone for alcohol dependent and hazardous drinking prisoners with HIV who are transitioning to the community. Contemp Clin Trials. 2014 Mar;37(2):209-18. doi: 10.1016/j.cct.2013.12.006. Epub 2013 Dec 31. PMID 24384538
- [Result] Vagenas P, Di Paola A, Herme M, Lincoln T, Skiest DJ, Altice FL, Springer SA. An evaluation of hepatic enzyme elevations among HIV-infected released prisoners enrolled in two randomized placebo-controlled trials of extended release naltrexone. J Subst Abuse Treat. 2014 Jul;47(1):35-40. doi: 10.1016/j.jsat.2014.02.008. Epub 2014 Mar 12. PMID 24674234
- [Result] Springer SA, Brown SE, Di Paola A, Altice FL. Correlates of retention on extended-release naltrexone among persons living with HIV infection transitioning to the community from the criminal justice system. Drug Alcohol Depend. 2015 Dec 1;157:158-65. doi: 10.1016/j.drugalcdep.2015.10.023. Epub 2015 Oct 28. PMID 26560326
- [Derived] Springer SA, Di Paola A, Barbour R, Azar MM, Altice FL. Extended-release Naltrexone Improves Viral Suppression Among Incarcerated Persons Living with HIV and Alcohol use Disorders Transitioning to the Community: Results From a Double-Blind, Placebo-Controlled Trial. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):92-100. doi: 10.1097/QAI.0000000000001759. PMID 29781884

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended-release Naltrexone: Subjects in this arm will receive monthly intramuscular gluteal injections of depot naltrexone 380mg (VIVITROL) for 6 months. The 1st injection will be administered prior to release from prison or jail.
  Vivitrol- Intramuscular naltrexone (depot-formulation): Subjects in this arm will receive monthly intramuscular gluteal injections of depot naltrexone 380mg (VIVITROL) for 6 months. The 1st injection will be administered prior to release from prison or jail.
Period: Overall Study
Arm/Group | Extended-release Naltrexone | Placebo
Started | 67 | 33
Completed | 67 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Naltrexone | Placebo | Total
Number analyzed (Participants) | 67 | 33 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 33 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (8.1) | 45.2 (8.9) | 45.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 21
  Male | 51 | 28 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 11 | 8 | 19
  Black (non Hispanic) | 46 | 19 | 65
  White (non Hispanic) | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 67 | 33 | 100
Alcohol use severity by AUDIT [Number; unit: participants]
  Abstinent or Low Risk Drinking | 2 | 0 | 2
  Hazardous Drinking | 5 | 2 | 7
  Harmful Drinking | 0 | 4 | 4
  Possible Dependence | 60 | 27 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Those Maintain or Improve to HIV RNA-1 Viral Load Less Then 400 Copies/mL
Description: Percentage of participants that maintained or improved a level of undetectable HIV viral load from baseline (closest viral load to time of release from incarceration) to 6 months post release. Missing lab values were considered to have a detectable HIV viral load.
Time Frame: Baseline to month 6 post release
Population: Logistic regression backward stepwise models were used to find predictors of HIV viral suppression.
Measure: Number; unit: percent of participants
Arm/Group | Intramuscular Naltrexone | Placebo
Number analyzed (Participants) | 67 | 33
percent of participants | 54 | 42

2. Secondary Outcome: Alcohol Treatment Outcome: Time to Alcohol Relapse
Description: Self reported time to first heavy drinking day after release from incarceration, up to 6 months
Time Frame: Post release
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Extended-release Naltrexone | Placebo
Number analyzed (Participants) | 67 | 33
days
  Age 20-29 | 24.1 (25.8) | 9.5 (10.6)
  Age 30-39 | 78.9 (49.5) | 73.9 (90.1)
  Agge 40-49 | 98.8 (70.4) | 85.0 (66.9)
  Age 50+ | 60.3 (74.1) | 64.1 (66.4)

3. Secondary Outcome: Alcohol Treatment Outcome: Change in Average Drinks Per Drinking Day
Description: The mean change from 12 weeks pre incarceration to 6 months post release from incarceration in average drinks per drinking day
Time Frame: 12 weeks prior to release from prison (baseline) to 6 months post release
Measure: Mean (Standard Deviation); unit: standard units of alcohol
Groups:
- Extended-release Naltrexone, Received 0-3 Injections: Subjects in this arm will receive monthly intramuscular gluteal injections of depot naltrexone 380mg (VIVITROL) for 6 months. The 1st injection will be administered prior to release from prison or jail.
  Vivitrol- Intramuscular naltrexone (depot-formulation): Subjects in this arm will receive monthly intramuscular gluteal injections of depot naltrexone 380mg (VIVITROL) for 6 months. The 1st injection will be administered prior to release from prison or jail.
- Placebo, Received 0-3 Injections: Subjects in this arm will receive monthly intramuscular gluteal injections of placebo for 6 months. The 1st injection will be administered prior to release from prison or jail.
  Placebo: Subjects in this arm will receive monthly intramuscular gluteal injections of placebo for 6 months. The 1st injection will be administered prior to release from prison or jail. Placebo will be provided by Alkermes pharmaceuticals, the manufacturer of VIVITROL. Placebo will be identical in shape and form to active drug.
Arm/Group | Extended-release Naltrexone, Received 0-3 Injections | Placebo, Received 0-3 Injections | Extended-release Naltrexone, Received 4-6 Injections | Placebo, Received 4-6 Injections
Number analyzed (Participants) | 40 | 19 | 27 | 14
standard units of alcohol | -16.6 (22.2) | -29.6 (27.5) | -17.4 (25.0) | -14.9 (16.3)

4. Secondary Outcome: Alcohol Treatment Outcome: Change in Percent of Heavy Drinking Days
Description: change in the percent of heavy drinking days from 12 weeks prior to incarceration to 6 months post release from incarceration.
Time Frame: change in percent of heavy drinking days12 weeks prior to release from prison (baseline), day of release, to 6 months post-release
Measure: Mean (Standard Deviation); unit: percent of heavy drinking days
Arm/Group | Extended-release Naltrexone, Received 0-3 Injections | Placebo, Received 0-3 Injections | Extended-release Naltrexone, Received 4-6 Injections | Placebo, Received 4-6 Injections
Number analyzed (Participants) | 40 | 19 | 27 | 14
percent of heavy drinking days | -38.3 (44.8) | -51.3 (41.1) | -63.6 (38.8) | -54.9 (46.9)

5. Other Pre Specified Outcome: Mean Change in CD4 Cell Count (Cells/mL)
Description: Baseline labs will be drawn while subjects is in prison, one to three months prior to release. Additionally, blood will be drawn every 3 months for 1 year to monitor changes in CD4 cell count.
Time Frame: Baseline and every 3 months for 1 year
Population: These data were not able to be collected for analysis.
Arm/Group | Extended-release Naltrexone, Received 0-3 Injections | Placebo, Received 0-3 Injections | Extended-release Naltrexone, Received 4-6 Injections | Placebo, Received 4-6 Injections
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: full study duration, up to 48 weeks post release
Arm/Group | Extended-release Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/33
Other Adverse Events (participants affected / at risk) | 9/67 | 2/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Naltrexone (N=67) | Placebo (N=33)
Nausea (Gastrointestinal disorders) | 9 (22) | 2 (4) — known medication side affect
headache (General disorders) | 5 (14) | 2 (3) — known drug side effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No